CLINICAL TRIAL: NCT02965768
Title: The Immune Effects of Low-dose Naltrexone in People With Myalgic Encephalopathy/Chronic Fatigue Syndrome (ME/CFS)
Brief Title: Immune Effects of Low-dose Naltrexone in ME/CFS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was temporarily suspended to focus on other projects, but was never resumed. No participants were determined eligible and none started the protocol.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jarred Younger, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: F160525003
Record Dates: First submitted 2016-11-14; First posted 2016-11-17 (Estimated); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Fatigue Syndrome, Chronic
MeSH Terms: conditions — Fatigue Syndrome, Chronic | interventions — Naltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind trial. An encrypted and password-protected database will contain (1) information about individual group assignment, and (2) blister pack codes (medication will be dispensed in blister packs by investigators based on these codes). An investigator not involved with data collection or participant interactions will randomly assign individuals to the treatment group and provide blister pack ID codes for each individual.
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDN arm (Active Comparator): Naltrexone HCl 4.5mg (standard-dose) or 3.0mg (optional-dose) x24 weeks
  Interventions: Drug: Naltrexone HCl
- Placebo/LDN arm (Other): Naltrexone HCl 4.5mg (standard-dose) or 3.0mg (optional-dose) Placebo
  Individuals will be switched between drugs as per approved schedule during the 24 weeks.
  Interventions: Drug: Naltrexone HCl

INTERVENTIONS:
Drug: Naltrexone HCl — 4.5 mg Naltrexone HCl, p.o., nocte (standard-dose); 3.0 mg Naltrexone HCl, p.o., nocte (optional-dose);
  Other Names: Low-dose Naltrexone; LDN

SUMMARY:
The main objective of this study is to test if naltrexone, when taken in low doses, has an anti-inflammatory effect that may be associated with positive clinical outcomes in people with chronic fatigue syndrome (CFS). In part, the present study, is a continuation of prior work in which we showed that chronic fatigue symptoms are associated with immune activity, and that low-dose naltrexone might exert anti-inflammatory effects in fibromyalgia, which is thought to share some pathophysiological and clinical characteristics with CFS.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the 1994 Case Definition criteria for CFS (assessed through semi-structured interview and the DePaul University Fatigue Questionnaire):

* Criteria:

  * Severe chronic fatigue ≥6 consecutive months not due to ongoing exertion or other medical condition associated with fatigue;
  * Fatigue interferes with daily activities and work;
  * Reports ≥4 symptoms that started with or after the fatigue, from:
* Post-exertion malaise >24 hours
* Unrefreshing sleep
* Short-term memory or concentration impairment
* Muscle pain
* Joint pain without swelling or redness
* Headaches of a new type/pattern/severity
* Lymph node tenderness
* Frequent or recurring sore throat 3. CFS symptoms for ≥12 months 4. Participant completes daily self-report during the 4-week baseline period; 5. Able to attend UAB on all scheduled appointments

Exclusion Criteria:

1. Blood draw contraindicated or otherwise not able to be performed
2. High-sensitivity c-reactive protein (HS-CRP) ≥3 mg/L
3. Erythrocyte sedimentation rate (ESR) >60 mm/hr
4. Positive rheumatoid factor
5. Positive anti-nuclear antibody (ANA)
6. Levels of thyroid stimulating hormone or free thyroxine outside UAB lab reference values
7. Diagnosed rheumatological or auto-immune condition
8. Clotting disorder
9. Use of blood thinning medication
10. Oral temperature >100˚F at baseline
11. Febrile illness or use of antibiotics in the 4 weeks before study commencement;
12. Planned surgery or procedures during the study period, or operated on in the 4 weeks before study commencement
13. Pregnant or planning on becoming pregnant within 6 months
14. Regular use of any anti-inflammatory medication (such as aspirin, ibuprofen, naproxen)
15. Known allergy or adverse effects following naltrexone or naloxone administration
16. Opioid use (self-reported or positive on urine test)
17. Significant psychological comorbidity that in the discretion of the investigator compromises study integrity and/or a baseline HADS depression subscale score of ≥16
18. Current litigation or worker's compensation claim
19. Current participation in another treatment trial
20. Vaccinated in the 4 weeks before study commencement (vaccination during the study period is allowed as long as the drug is administered at least 4 weeks prior to a study blood draw).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2022-08-25 (Actual); Study Completion 2022-08-25 (Actual)

PRIMARY OUTCOMES:
Reduction in plasma inflammatory biomarkers | Four-week baseline; 12 weeks drug
  Levels of plasma IL-1B, TNFa, IL6, IL12, and IL17 will be tested as the primary biomarkers of interest.

SECONDARY OUTCOMES:
Durability of reduction in plasma inflammatory biomarkers | Baseline; 12 weeks drug; 24 weeks drug
  Levels of plasma IL-1B, TNFa, IL6, IL12, and IL17 will be tested as the primary biomarkers of interest. 24 weeks vs 12 weeks drug.
Reduction in self-reported fatigue | 12 weeks drug
  Fatigue will be reported daily on a hand-held computer device.
Increase in physical function | 12 weeks drug
  Physical function will be reported weekly on a Patient-Specific Functional Scale.
Reduction in self-reported symptoms of (i) depression, (ii) anxiety | 12 weeks drug
  Symptoms of depression and anxiety will be reported weekly on a Hospital Anxiety and Depression Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Jarred Younger, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Younger J, Parkitny L, McLain D. The use of low-dose naltrexone (LDN) as a novel anti-inflammatory treatment for chronic pain. Clin Rheumatol. 2014 Apr;33(4):451-9. doi: 10.1007/s10067-014-2517-2. Epub 2014 Feb 15. PMID 24526250